CLINICAL TRIAL: NCT01408550
Title: NPB-01(Intravenous Immunoglobulin) Therapy for Patients With Bullous Pemphigoid Unresponsive to Corticosteroids: Randomized, Double-Blind, Placebo Control,Parallel Assignment Study(Phase III)
Brief Title: Phase III Clinical Trial of NPB-01 in Patients With Bullous Pemphigoid Unresponsive to Corticosteroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Nihon Pharmaceutical Co., Ltd, Clinical Development Department
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPB-01-06/C-01
Record Dates: First submitted 2011-07-27; First posted 2011-08-03 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Bullous Pemphigoid
Keywords: IVIG in pemphigoid; Patients with bullous pemphigoid unresponsive to corticosteroids
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPB-01 (Active Comparator): Active Comparator: 1 Intravenous immunoglobulin
  Interventions: Drug: NPB-01
- Placebo (Placebo Comparator): Placebo Comparator: 2 Physiological saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NPB-01 — Intravenous immunoglobulin
  Arms: NPB-01
Drug: Placebo — Physiological saline
  Arms: Placebo

SUMMARY:
Patients diagnosed with bullous pemphigoid were confirmed based on the investigators national diagnostic criteria. Patients who meet all inclusion criteria and do not conflict with the exclusion criteria will receive NPB-01 (intravenous immunoglobulin) 400mg/kg/day for five consecutive days or Placebo(physiological saline). Subsequently, efficacy of NPB-01 for therapy of bullous pemphigoid will be evaluated the score using pemphigus disease area index (PDAI) and pemphigoid activity score involving skin lesion area and Number of new blisters.

As a safety endpoint, the safety of NPB-01 will be investigated the occurrence of adverse events by 57 days after the start of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with corticosteroids over 0.4mg/kg/day(Prednisolone) at informed consent.
2. Patients with continued treatment for bullous pemphigoid without add or change the treatment after informed consent.
3. Patients who the score using Pemphigus Disease Area Index(PDAI) is score10 and more before study medication received.
4. Patients who the score using Pemphigus Disease Area Index(PDAI) is not improve before study medication received.
5. Patients with twenty years old at informed consent.
6. Patients with hospitalization during five consecutive days of study medication and seven consecutive days after administration of study medication .

Exclusion Criteria:

1. Patients treated with plasmapheresis at 28 days before informed consent.
2. Patients treated with corticosteroids pulse therapy(methylprednisolone over 0.5g/day) at 14 days before informed consent.
3. Patients treated with intravenous immunoglobulin at 56 days before informed consent.
4. Patients who receive or adjust in increments immunosuppressants at 14 days before informed consent.
5. Patients with malignancy or a history of this disease.
6. Patients with history of shock for NPB-01.
7. Patients with history of hypersensitivity for NPB-01.
8. Patients with IgA deficiency.
9. Patients with impaired liver function.
10. Patients with impaired renal function.
11. Patients with cerebro- or cardiovascular disorders.
12. Patients with high risk of thromboembolism.
13. Patients with hemolytic/hemorrhagic anemia.
14. Patients with decreased cardiac function.
15. Patients with decreased platelet.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The score using Pemphigus Disease Area Index (PDAI) | 15 days

SECONDARY OUTCOMES:
Pemphigoid Activity Score | 8 weeks
anti-BP180 antibody titers | 8 weeks
Oral Steroid dose | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka, Japan